CLINICAL TRIAL: NCT02553850
Title: A SURVEY TO STUDY THE CORRELATION BETWEEN THE SERUM LEVELS OF BONE TURNOVER MARKERS AND THE CLINICAL PICTURE IN PATIENTS WITH BREAST CANCER AND BONE METASTASES RECEIVING IBRADONIC ACID TREATMENT
Brief Title: An Observational Study in Patients With Breast Cancer and Bone Metastases Receiving Ibandronate (Bondronat)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML20416
Record Dates: First submitted 2015-09-08; First posted 2015-09-18 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Ibandronate: Patients receiving ibandronate will be evaluated for bone turnover markers for 12 months. Ibandronate is not an investigational medicinal product (IMP) in this study.

SUMMARY:
This open non-randomized, single-arm, multicenter, observational study is designed to evaluate the correlation between bone turnover markers and the response to treatment in patients with breast cancer and bone metastases. In this observational study, ibandronate (Bondronat) will be prescribed and used in accordance with the standards of care. Data will be collected for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All criteria in accordance with the Summary of Product Characteristics of Bondronat (ibandronate)
* Adult patients greater than (>) 18 years of age
* Histologically confirmed breast cancer
* Confirmed bone metastasis (by bone scintigraphy, X-ray, computed tomography or magnetic resonance imaging)
* Life expectancy >6 months
* No previous bisphosphonate therapy
* Patients signed written informed consent form before study start

Exclusion Criteria:

* All criteria in accordance with the Summary of Product Characteristics of Bondronat(ibandronate)
* Hypersensitivity to the active substance or any of the excipients of Bondronat (ibandronate)
* Hypersensitivity to bisphosphonates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer and bone metastases who have been prescribed ibandronate (Bondronat) will be evaluated in the routine oncological setting for 12 months.
Sampling Method: Probability Sample
Enrollment: 442 (Actual)
Dates: Start 2007-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Beta C-terminal telopeptide (B-CTx) level | 12 months
Treatment response rate | 12 months

SECONDARY OUTCOMES:
Number of patients who died due to progression of breast cancer | 12 months
Safety: Incidence of adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- Hungary (15):
  - Budapest
  - Debrecen
  - Győr
  - Gyula
  - Kaposvár
  - Nyíregyháza
  - Pécs
  - Szeged
  - Szekszárd
  - Székesfehérvár
  - Szolnok
  - Szombathely
  - Tatabánya
  - Veszprém
  - Zalaegerszeg-Pozva